CLINICAL TRIAL: NCT02569645
Title: Phase 2 Trial of Rosuvastatin (Crestor®) Combined With Standard Chemoradiation Therapy in the Treatment of High-Risk Locally Advanced Rectal Cancer
Brief Title: Rosuvastatin in the Treatment of Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-064
Record Dates: First submitted 2015-09-24; First posted 2015-10-07 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Rosuvastatin
MeSH Terms: conditions — Rectal Neoplasms | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm - Rosuvastatin (Experimental): This is a single arm, of Rosuvastatin (Crestor®) 40 mg orally daily starting 2 weeks prior to the initiation of radiation at week 1 and stopped 4 weeks after the completion of radiation at the start of week 12 or 13, depending on whether 25 or 30 fractions of radiotherapy are given.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 40 mg rosuvastatin orally once per day with or without food, swallowed whole (not chewed, crushed or divided) starting 2 weeks prior to the initiation of radiation therapy and stopped at 4 weeks after the completion of radiation. Total duration of Rosuvastatin is 11 weeks if 25 fractions of radiotherapy are given, or 12 weeks if 30 fractions of radiotherapy are given.
  Other Names: Crestor

SUMMARY:
This study will evaluate whether the addition of Rosuvastatin to standard chemoradiation therapy for the treatment of locally advanced rectal cancer may improve the pathological response rate and survival compared to standard chemoradiation therapy alone.

DETAILED DESCRIPTION:
The standard treatment of locally advanced rectal cancer involves neoadjuvant chemoradiation therapy (CRT) followed by surgery and further adjuvant chemotherapy. The pathologic complete responses associated with neoadjuvant CRT are 10-20%. The prognosis of patients undergoing neoadjuvant CRT is associated to the extent of post-treatment tumour regression, the final primary tumour stage and presence of involved lymph nodes in the surgical specimen. This data suggests that treatments that enhance the pathological response may result in improvements in survival.

Overwhelming preclinical and clinical evidence suggests that statins demonstrate anticancer properties and sensitize cancer tissues and protects normal tissues to the effects of radiation. Hence, the investigators hypothesize that the addition of rosuvastatin to standard CRT for the treatment of locally advanced rectal cancer may improve the pathological response rate. This protocol describes an open-label single-arm phase 2 study designed to test this hypothesis. Moreover, this study will also identify genetic, serological, and pathological biomarkers that may be both prognostic and predictive of response and toxicity to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical stage 2-3 rectal adenocarcinoma, cT3/4N0/M0 or Tx N1-2/M0, within 5 cm of anal verge or less than 12cm from anal verge and threatened circumferential resection margin (≤3mm). Patients must have histological confirmation of rectal adenocarcinoma prior to registration.
2. Patients must be 18 years or older.
3. Able to swallow oral medication.
4. Previous surgery, not for primary treatment of current rectal cancer, is permitted provided that wound healing has occurred and at least 14 days have elapsed prior to registration if surgery was major.
5. ECOG 2 or less.
6. Laboratory Requirements (must be done within 7 days prior to registration):

   a. Hematology: i. Hemoglobin ≥90 g/L ii. Granulocytes (AGC) ≥ 1.5 x 109/L iii. Platelets ≥ 100 x 109/L b. Chemistry: i. Bilirubin ≤1.5 x UNL ii. ALT or AST ≤ 1.5 x UNL iii. Proteinuria ≤ grade 1 iv. Thyroid function within normal limits (TSH or free T4 within normal limits after correction) v. CPKs ≤ ULN, vi. Urinary myoglobin within normal limits Note: If serum creatinine is abnormal, a creatinine clearance should be calculated and be ≥ 60 ml/min.
7. Women must be post-menopausal, surgically sterile or use two reliable forms of contraception if of child-bearing potential. Women of childbearing potential must have a urine pregnancy test taken and proven negative within 7 days prior to registration. Men must be surgically sterile or use an effective barrier method of contraception if sexually active with a woman of child-bearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose.
8. Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. It will be the responsibility of the local participating investigators to obtain the necessary local clearance. The patient must sign the consent form prior to registration. The consent form for this study must contain a statement, which gives permission for the sponsor and monitoring agencies to review patient records.
9. Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 1⁄2 hours driving distance) placed on patients being considered for this trial. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.

Exclusion Criteria:

1. Patients of Asian ethnicity (having Filipino, Chinese, Japanese, Korean, Vietnamese, or South Asian origin) will be excluded due to increased risk of toxicity.
2. Previous and concurrent, experimental, chemotherapy, or radiotherapy treatment for primary rectal carcinoma.
3. Statin exposure in the last 5 years.
4. Known evidence of distant metastatic disease on staging investigation, including a CT of the chest, abdomen, and pelvis performed within 6 weeks prior to registration.
5. Known history of previous malignancy, except adequately treated non-melanoma skin cancer or other solid tumour treated curatively with no evidence of disease for >5 years.
6. Patients with malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease significantly affecting gastrointestinal (GI) function.
7. Patients with a known history of documented upper GI bleeding or upper GI ulcerative disease.
8. Patients with hyperlipidemia with clinical indication for statin therapy or other prescribed medication (determination of acceptable fasting lipid values should be in accordance with current dyslipidemia management guidelines).
9. Patients with inadequately treated hypothyroidism, as determined by the investigator.
10. Patients with a known history of myopathy or rhabdomyolysis.
11. Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction.
12. Deemed by the physician to be at low risk for recurrence.
13. No other non-malignant systemic disease that would preclude rosuvastatin administration or prolonged follow-up.
14. Concurrent chronic use of NSAIDs.
15. Concurrent chronic drug therapy with cyclosporine, colchicine, coumarin anticoagulants, amiodarone, gemfibrozil, other lipid-lowering therapies (e.g., fibrates or niacin), lopinavir/ritonavir, azole antifungals, and macrolide antibiotics.
16. Known personal or family history of hereditary neuromuscular disorders.
17. Known previous history of muscular toxicity with another HMG-CoA reductase inhibitor.
18. Known history of alcohol abuse.
19. Any known condition that could affect absorption of study oral drugs (capecitabine and rosuvastatin).
20. Known contraindication to statin.
21. Pregnant or nursing.
22. Patients with symptomatic inflammatory bowel disease.
23. Patients with uncontrolled hypothyroidism.
24. Patients with chronic liver or disease.
25. Patients with unexplained elevated serum transaminases exceeding 3x ULN.
26. Patients known to be suffering from infection with HIV, Tuberculosis, Hepatitis C or Hepatitis B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-11; Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
To determine the pathological complete response rate in patients with high-risk locally advanced rectal cancer treated with standard neo-adjuvant chemotherapy and radiation in combination with rosuvastatin. | Up to 3 years
  The rate of post-surgical specimens that demonstrate absence of any residual invasive disease or Grade 4 (complete) histological regression using the Dworak classification.

SECONDARY OUTCOMES:
To determine the Ro resection rate | Up to 3 years
  The rate that the surgical margins are negative of any invasive disease.
To determine the pathological near-complete or complete tumour response rate | Up to 3 years
  Grade 3 (near-complete) or 4 (complete) histological regression using the Dworak classification.
To determine the sphincter preservation rate | Up to 3 years
  The proportion of patients that undergo a sphincter preservation surgery versus abdominoperineal resection.
To determine the down staging rate | Up to 3 years
  Proportion of patients that have a down staging of the primary tumour and/or lymph nodes; i.e. comparison between cT/N and ypT/N
To determine 3-year disease free survival | Up to 3 years
  The proportion of patients alive with no clinical, radiological, or pathological evidence of rectal cancer recurrence at 3 years, starting at the time treatment was initiated. This definition includes, recurrence or relapse of rectal cancers, second primary cancer or death as events
To determine 3-year overall survival | Up to 3 years
  The proportion of patients alive at 3 years, starting at the time treatment was initiated.
To determine the neoadjuvant rectal cancer (NAR) score | Up to 3 years
  A surrogate endpoint of overall survival following neoadjuvant rectal cancer therapy.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | Up to 3 years
To identify the genetic biomarkers that may be both prognostic and predictive of response and toxicity to treatment. | up to 3 years
  BRAF and KRAS genetic testing. Direct exon sequencing.
To identify serological biomarkers that may be both prognostic and predictive of response and toxicity to treatment. | up to 3 years
  Changes in the levels of HMG CoA reductase pathway metabolites (Mevalonate, Ubiquinone) will also be performed using pre- and post-treatment serological markers.
To identify pathological biomarkers that may be both prognostic and predictive of response and toxicity to treatment. | up to 3 years
  IHC using pre- and post FFPE tumour tissue samples. (Ki67, phopsorylated AKT, HMG CoA reductase, GGPS1 and ApopTag, p21, p27 and rhoA)
Tmax will be collected as pharmacokinetic data | up to 3 years
Cmax will be collected as pharmacokinetic data | up to 3 years
T1/2 will be collected as pharmacokinetic data | up to 3 years
Dose normalized Cmax will be collected as pharmacokinetic data | up to 3 years
Area under the curve (AUC) will be collected as pharmacokinetic data | up to 3 years
Dose normalized AUC will be collected as pharmacokinetic data | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jose Monzon, PhD MD FRCPC, Principal Investigator — Tom Baker Cancer Centre
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided